CLINICAL TRIAL: NCT01884467
Title: Randomized Placebo-Controlled Trial of Gentamicin Bladder Instillation for the Prevention of Urinary Tract Infection in Adults at High Risk for Cystitis Due to Intermittent Catheterization
Brief Title: Gentamicin Bladder Instillation Trial
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gillette Children's Specialty Healthcare (Other)
Responsible Party: Principal Investigator, Sean P. Elliott, M.D., M.S., Associate Professor and Vice Chair, Director of Reconstructive Urology, University of Minnesota, Gillette Children's Specialty Healthcare
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 1210M21603
Record Dates: First submitted 2013-06-18; First posted 2013-06-24 (Estimated); Last update posted 2015-04-09 (Estimated); Status verified 2015-04

CONDITIONS: Urinary Tract Infections
Keywords: Urinary Tract Infections; Gentamicin
MeSH Terms: conditions — Urinary Tract Infections | interventions — Gentamicins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gentamicin (Experimental): Intervention: Gentamicin; Dosage form: 120mg reconstituted in 250cc of normal saline; Dosage: 30mL; Frequency: nightly instillation into bladder (to remain overnight until draining it out in morning); Duration: 1 year
  Interventions: Drug: Gentamicin
- Placebo (Placebo Comparator): Drug: Normal saline; Dosage form: N/A; Dosage: 30 mL; Frequency: nightly bladder instillation; Duration: 1 year
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Gentamicin — Comparison of Gentamicin versus placebo
  Other Names: Garamycin solution
  Arms: Gentamicin
Drug: Placebo
  Arms: Placebo

SUMMARY:
Recurrent UTIs are common among patients on IC. These create significant patient morbidity and healthcare burden. In desperation, many physicians prescribe prophylactic oral or intravesical antibiotics. This practice is common among our Gillette clinic patients. However, the benefit is unclear and the risks are not insignificant. As such, practice variation is significant. In order to better define the evidence for or against gentamicin bladder irrigation and thus inform clinical practice both locally at our Gillette urology clinic and for practitioners at large we will pursue the following specific aims:

1. Compare rates of symptomatic urinary tract infection and asymptomatic bacteriuria among a population of Gillette patients on IC with and without gentamicin bladder instillation.
2. Compare antibiotic resistance rates among a population of Gillette patients on IC with and without gentamicin bladder instillation.

DETAILED DESCRIPTION:
In the Gillette Lifetime Urology clinic, gentamicin bladder instillation (GBI) for UTI prophylaxis is common practice among our neurogenic bladder patients in IC. However, as previously shown, the evidence supporting this practice is mixed. Potential risks of this practice include wasted costs, wasted materials, wasted time and growing antibiotic resistance. Potential benefits include reduced use of systemic antibiotics, a reduction in symptomatic UTIs and fewer hospitalizations for febrile UTIs. We seek to define the evidence for or against this practice by completing a double-blind randomized controlled trial of GBI vs. NS instillation. Such a trial would benefit our Gillette patients and the community of patients on IC worldwide.

Recurrent UTIs are common among patients on IC. These create significant patient morbidity and healthcare burden. In desperation, many physicians prescribe prophylactic oral or intravesical antibiotics. This practice is common among our Gillette clinic patients. However, the benefit is unclear and the risks are not insignificant. As such, practice variation is significant. In order to better define the evidence for or against gentamicin bladder irrigation and thus inform clinical practice both locally at our Gillette urology clinic and for practitioners at large we will pursue the following specific aims:

1. Compare rates of symptomatic urinary tract infection and asymptomatic bacteriuria among a population of Gillette patients on IC with and without gentamicin bladder instillation.
2. Compare antibiotic resistance rates among a population of Gillette patients on IC with and without gentamicin bladder instillation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients (>=16 years of age) with any diagnosis on IC of the bladder.
2. Patients may catheterize either thru the urethra or a stoma (e.g. Mitrofanoff).
3. A history of recurrent symptomatic UTI's (at least 3 per year).
4. Patient must be able to travel to Gillette's Lifetime clinic for quarterly urine cultures
5. Patient must have an "informed other" that can supplement any missing study information (incident UTI, treatment information, etc.)

Exclusion Criteria:

1. Patients currently on oral or intravesical antibiotic prophylaxis refusing to or not able to discontinue prophylaxis.
2. Patients colonized with gentamicin-resistant bacteria on baseline urine culture or a gentamicin allergy.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2013-05; Primary Completion 2015-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Symptomatic UTI | one year
  Our primary outcome will be febrile or symptomatic UTI, defined as fever or abdominal pain or new bladder symptoms such as pain, urinary incontinence, hematuria or more frequent bladder spasms plus urine culture demonstrating >103 CFUs of a single dominant bacteria or >105 of multiple bacteria.

SECONDARY OUTCOMES:
Asymptomatic UTI | one year
  A quarterly urine culture will be performed at Gillette's Lifetime Clinic to assess asymptomatic bacteriuria. Asymptomatic bacteriuria will be defined as an asymptomatic patient with urine sample culture positive for typical bacteria.

CONTACTS AND LOCATIONS:
Overall Officials: Sean P Elliott, MD, MS, FACS, Principal Investigator — Gillette Children's Specialty Healthcare
Locations (1):
- Gillette Lifetime Specialty Healthcare, Saint Paul, Minnesota, United States